CLINICAL TRIAL: NCT02088450
Title: Systolic Hypertension in Europe Trial
Brief Title: Systolic Hypertension in Europe Placebo-Controlled Trial
Acronym: Syst-Eur
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Syst-Eur
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Isolated Systolic Hypertension
Keywords: Cardiovascular complications; Clinical trial; Elderly; Isolated systolic hypertension; Stroke
MeSH Terms: conditions — Isolated Systolic Hypertension; Stroke | interventions — Nitrendipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment (Active Comparator): Active treatment with nitrendipine (10-40 mg/day). If necessary, the dihydropyridine calcium-channel blocker was combined with or replaced by enalapril maleate (5-20 mg/day), hydrochlorothiazide (12.5-25 mg/day), or both drugs.
  Interventions: Drug: Active treatment with nitrendipine (10-40 mg/day).
- Placebo (Placebo Comparator): Placebo tablets were identical to the study drugs with a similar schedule.
  Interventions: Drug: Active treatment with nitrendipine (10-40 mg/day).

INTERVENTIONS:
Drug: Active treatment with nitrendipine (10-40 mg/day). — If necessary, the dihydropyridine calcium-channel blocker was combined with or replaced by enalapril maleate (5-20 mg/day), hydrochlorothiazide (12.5-25 mg/day), or both drugs.

SUMMARY:
The Syst-Eur Trial is a concerted action of the European Community's Medical and Health Research Programme. The trial is carried out in consultation with the World Health Organization, the International Society of Hypertension, the European Society of Hypertension and the World Hypertension League. Syst-Eur is a multicentre trial designed by the European Working Party on High Blood Pressure in the Elderly (EWPHE), to test the hypothesis that antihypertensive treatment of elderly patients with isolated systolic hypertension results in a significant change in stroke morbidity and mortality. Secondary endpoints include cardiovascular events, such as myocardial infarction and congestive heart failure. To be eligible patients must be at least 60 years old and have a systolic blood pressure averaging 160-219 mmHg with a diastolic pressure less than 95 mmHg. Patients must give their informed consent and be free of major cardiovascular and non-cardiovascular diseases at entry. The patients are randomized to active treatment or placebo. Active treatment consists of nitrendipine (10-40 mg/day), combined with enalapril (5-20 mg/day) and hydrochlorothiazide (12.5-25 mg/day), as necessary. The patients of the control group receive matching placebos. The drugs (or matching placebos) are stepwise titrated and combined in order to reduce systolic blood pressure by 20 mmHg at least to a level below 150 mmHg. Morbidity and mortality are monitored to enable an intention-to-treat and per-protocol comparison of the outcome in the 2 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years old.
* Sitting systolic blood pressure on masked placebo, during run-in phase of 160 to 219 mmHg, with a sitting diastolic blood pressure below 95 mmHg and a standing systolic blood pressure of at least 140 mmHg
* Informed consent must be obtained

Exclusion Criteria:

* Systolic hypertension is secondary to a disorder that needed specific medical or surgical treatment.
* Retinal haemorrhage or papilloedema;
* Congestive heart failure
* Dissecting aortic aneurysm
* Serum creatinine concentration at presentation of 180µmol/L or more.
* History of severe nose bleeds.
* Stroke or myocardial infarction in the year before the study.
* Dementia.
* Substance abuse.
* Any disorder prohibiting a sitting or standing position.
* Any severe concomitant cardiovascular or non-cardiovascular disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4695 (Actual)
Dates: Start 1990-02; Primary Completion 1997-02 (Actual); Study Completion 1997-02 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke | 3-monthly visits up to 5 years
  Available in Lancet 1997; 350:757-764

SECONDARY OUTCOMES:
Death | 3-monthly visits up to 5 years
  Available in Lancet 1997; 350:757-764
Myocardial infarction | 3-monthly visits up to 5 years
  Available in Lancet 1997; 350:757-764
Congestive heart failure | 3-monthly visits up to 5 years
  Available in Lancet 1997; 350:757-764

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Staessen, MD, PhD, Principal Investigator — University of Leuven

IPD SHARING:
Plan to Share IPD: Yes
Syst-Eur data are available on request by other investigators, whose research is ethically approved.

REFERENCES:
- [Derived] Grobman B, Turkson-Ocran RN, Staessen JA, Yu YL, Lipsitz LA, Mukamal KJ, Juraschek SP. Body Position and Orthostatic Hypotension in Hypertensive Adults: Results from the Syst-Eur Trial. Hypertension. 2023 Apr;80(4):820-827. doi: 10.1161/HYPERTENSIONAHA.122.20602. Epub 2023 Feb 6. PMID 36744469
- [Derived] Hara A, Thijs L, Asayama K, Jacobs L, Wang JG, Staessen JA. Randomised double-blind comparison of placebo and active drugs for effects on risks associated with blood pressure variability in the Systolic Hypertension in Europe trial. PLoS One. 2014 Aug 4;9(8):e103169. doi: 10.1371/journal.pone.0103169. eCollection 2014. PMID 25090617